CLINICAL TRIAL: NCT05012345
Title: Distal Radial Fractures in Adult Patients: 4 Weeks Versus 6 Weeks of Cast Immobilization Following Closed Reduction.
Brief Title: Distal Radial Fractures in Adult Patients: 4 Weeks Versus 6 Weeks of Cast Immobilisation Following Closed Reduction.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cork University Hospital (Other)
Responsible Party: Principal Investigator, Hany Elbardesy, Principal Investigator, Cork University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ECM 3 (vvv) 09/02/2021
Record Dates: First submitted 2021-07-24; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Distal Radius Fracture
Keywords: distal radius fracture, 4 weeks, 6 weeks.
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: A prospective single-blinded randomised clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Data from the demographic data collection and the outcome parameters will be cleaned blindly from the treatment data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4 Weeks cast immobilisation (Experimental): Patients with fracture distal radius ( indicated for conservative treatment) will stay in a below-elbow cast for 4 weeks. Following immobilisation, treatment will be the same for both groups, in which additional physiotherapy after removal of the cast is advised and exercises to train wrist function will be given. As extra structured advice programmes may cause no extra benefit for the patient, this was not generally prescribed. However, during FU visits, patients will be asked if they were treated by a physiotherapist. If this is the case, details on the number of sessions per week and the total number of weeks the patient received physiotherapy, will be collected.
  Interventions: Procedure: Below Elbow cast
- 6 Weeks cast immobilisation (Experimental): Patients with fracture distal radius ( indicated for conservative treatment) will stay in a below-elbow cast for 6 weeks. Following immobilisation, treatment will be the same for both groups, in which additional physiotherapy after removal of the cast is advised and exercises to train wrist function will be given. As extra structured advice programmes may cause no extra benefit for the patient, this was not generally prescribed. However, during FU visits, patients will be asked if they were treated by a physiotherapist. If this is the case, details on the number of sessions per week and the total number of weeks the patient received physiotherapy, will be collected.
  Interventions: Procedure: Below Elbow cast

INTERVENTIONS:
Procedure: Below Elbow cast — below-elbow cast ( 4 or 6 weeks )

SUMMARY:
A single-blinded randomized controlled trial is initiated. Four weeks of plaster cast immobilization is compared with six weeks of plaster cast immobilization in adult patients with adequately reduced distal radius fracture. Primary outcome parameters are functional outcomes measured with the Patient Rated Wrist Evaluation after 6 months of follow-up (FU). Secondary outcomes are Disability of Arm, Shoulder and Hand Score after 6 months and one year, 36-Item Short-Form Health Survey after 6 months and one year, functional outcome earlier in Follow up (6 weeks, 12 weeks, 6 months, and one year), range of motion, pain level, and complications: number of re-interventions, secondary displacement, delayed and non-union.

DETAILED DESCRIPTION:
This study will be conducted as a prospective single-blinded randomized clinical trial in a level one trauma center serving the southeast of Ireland. In this study, 4 weeks of plaster immobilization will be compared with 6 weeks of plaster immobilization. The methods of this study protocol are comparable to a previously published article comparing 3 weeks of cast immobilization to 5 weeks of cast immobilization in adult patients with non-displaced distal radius fractures. Patients will be treated in a lower arm cast in a neutral position. Following immobilization, treatment will be the same for both groups, in which additional physiotherapy after removal of the cast is advised, and exercises to train wrist function will be given. As extra structured advice programs may cause no extra benefit for the patient, this was not generally prescribed. However, during follow-up visits, patients will be asked if they were treated by a physiotherapist. If this is the case, details on the number of sessions per week and the total number of weeks the patient received physiotherapy, will be collected.

Patients will only be able to participate if closed reduction of the DRF is adequate. The indication for reduction will be set, using the Lidström criteria for misalignment. Patients will only be able to participate in this study if reduction is performed successfully. Successful reduction will be classified as radial shortening <3 mm, dorsal tilt <10° or intra-articular step-off <2 mm, according to the guidelines of the American Academy of Orthopaedic Surgeons.

After providing informed consent, eligible patients will be randomised after 2 weeks when the fracture has proven to be stable. An independent research assistant will perform concealed permuted block randomisation using a computer-generated randomisation schedule after stratification for fracture type, gender, and age. Allocation will be at random in four blocks. To prevent bias, stratification by age (younger and older than 60 years) and gender will be performed . Randomisation between another 2 or 4 weeks cast immobilisation will be performed to complete a total of 4 and 6 weeks of cast immobilisation, respectively. Randomisation will occur after informed consent.

cast removal, number of re-interventions, delayed and non-unions and Complex regional Pain Syndrome (CRPS).

At each FU visit, the research coordinator or research assistant will ascertain patient status (ie, secondary interventions, adverse events/complications, deaths) and will verify the information within medical records. All adverse events will be addressed to the principal investigator. At each FU visit, the patients will be asked to indicate the actual pain level on a VAS. Patients will also be asked if they have any complaints of their treatment and will be asked if they are currently treated by a physical therapist. At each visit from 8 weeks onwards, the range of motion of the wrist will be measured using a goniometer, according to the reference values for joint range of motion published by the American Academy of Orthopaedic Surgeons. In addition, patients will be asked to complete the questionnaires relating to disability. Plain X-rays of the wrist will be made at the time of presentation in the hospital (ED), after 1 and 2 weeks, 4 or 6 weeks, and at the follow-up visit after 8 weeks, 3 months, 6 months, and one year. The X-ray at 6 months will be taken in order to determine the grade of degenerative joint changes. The time to define the presence of a delayed- or non-union will be at 3 or 6 months. The sample size of 44 patients per treatment group is calculated with a power (1-β) of 80% and a type I error (α) of 5%, allowing for 10% dropout. In this study, we decided to include 50 patients per treatment group. To allow a 10% dropout in this study, in total 100 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

1. Primary displaced distal radius fracture
2. age older than 18 years.
3. Adequate closed reduction of the distal radius fracture according to Lidström criteria for misalignment.

Exclusion Criteria:

1. Ipsilateral fractures proximal to the distal radius.
2. Pre-existent abnormalities or functional deficits of the fractured wrist that influences the patient reported function of the wrist.
3. Open fractures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-20 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Patient Rated Wrist Evaluation (PRWE) | One year
  is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living
Patient Rated Wrist Evaluation (PRWE) | Three months
  is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living
Patient Rated Wrist Evaluation (PRWE) | Six months
  is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living
Quick Disability of Arm and Shoulder (DASH) | 3 months
  is a self-report questionnaire that assesses a person's perceived level of incapacity pertaining to disability of the arm, shoulder, and hand and is based on the 30-item DASH instrument, where each item on the QuickDASH was retained relative to key concepts of upper-limb functioning as well as the selection of the highest ranked items from the original according to their psychometric properties
Quick Disability of Arm and Shoulder (DASH) | 6 months
  is a self-report questionnaire that assesses a person's perceived level of incapacity pertaining to disability of the arm, shoulder, and hand and is based on the 30-item DASH instrument, where each item on the QuickDASH was retained relative to key concepts of upper-limb functioning as well as the selection of the highest ranked items from the original according to their psychometric properties
Quick Disability of Arm and Shoulder (DASH) | One year
  is a self-report questionnaire that assesses a person's perceived level of incapacity pertaining to disability of the arm, shoulder, and hand and is based on the 30-item DASH instrument, where each item on the QuickDASH was retained relative to key concepts of upper-limb functioning as well as the selection of the highest ranked items from the original according to their psychometric properties

SECONDARY OUTCOMES:
Range of Movement | 3 months
  Flexion, Extension, radial and ulnar deviation
Range of Movement | 6 months
  Flexion, Extension, radial and ulnar deviation
Range of Movement | one year
  Flexion, Extension, radial and ulnar deviation
Complications | one year
  Stiffness, delayed and non-union and complex regional pain syndrome (CRPS).

CONTACTS AND LOCATIONS:
Locations (1):
- Cork University Hospital, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: July 2022

REFERENCES:
- [Derived] Elbardesy H, Yousaf MI, Reidy D, Ansari MI, Harty J. Distal radial fractures in adults: 4 versus 6 weeks of cast immobilisation after closed reduction, a randomised controlled trial. Eur J Orthop Surg Traumatol. 2023 Dec;33(8):3469-3474. doi: 10.1007/s00590-023-03574-2. Epub 2023 May 16. PMID 37191887